CLINICAL TRIAL: NCT04711395
Title: The Application of Lens Dysfunction Index (DLI) in the Timing of Age-related Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Deputy Dean, Wenzhou Medical University
Other Study IDs: YZhao
Record Dates: First submitted 2021-01-05; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Age-Related Cataract
Keywords: Age-related cataract; DLI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cataract Surgery Group
  Interventions: Device: measure the preoperative DLI、 SS-OCT image of the lens,、take photos of the anterior segment and self-scoring of the preoperative visual quality assessment scale.
- Non-surgical group
  Interventions: Device: measure the preoperative DLI、 SS-OCT image of the lens,、take photos of the anterior segment and self-scoring of the preoperative visual quality assessment scale.

INTERVENTIONS:
Device: measure the preoperative DLI、 SS-OCT image of the lens,、take photos of the anterior segment and self-scoring of the preoperative visual quality assessment scale. — subjects in the observation group and Healthy used iTrace ocular aberration analyzer（itracey Technologies）and IOL-Master 700 biometer to measure the preoperative DLI(Dysfunctional lens index) and SS-OCT image of the lens, and The researchers used the anterior segment slit lamp to take photos of the anterior segment of the subject's lens in a state of dilated pupils .and self-scoring of the preoperative visual quality assessment scale.

SUMMARY:
Before cataract surgery, subjects in the observation group used iTrace ocular aberration analyzer（itracey Technologies）and IOL-Master 700 biometer to measure the preoperative DLI(Dysfunctional lens index) and SS-OCT image of the lens, and The researchers used the anterior segment slit lamp to take photos of the anterior segment of the subject's lens in a state of dilated pupils .and self-scoring of the preoperative visual quality assessment scale. Healthy subjects in the control group also need to complete the above inspections. After that, three experienced cataract specialist surgeons combined the preoperative optometry data of each subject, the photos of the LOCS III anterior segment and the Catquest-9SF questionnaire score to determine whether each subjects should undergo cataract surgery. The subjects were divided into cataract surgery group and non-surgical group. Finally, statistically study the correlation between the DLI index and the degree of lens opacity that has been collected, and use the ROC curve to calculate the DLI as the best cut-off point of DLI to distinguish whether to perform cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years old
* Healthy volunteers with no history of systemic or ocular diseases
* patients with simple age-related cataracts without other ocular diseases
* those who can communicate with the tester at a normal level
* those who can express their own ideas independently

Exclusion Criteria:

* irregular corneal astigmatism
* corneal opacity
* corneal scars
* corneal dystrophy
* shallow of anterior chamber
* retinal abnormalities
* history of eye surgery or laser treatment
* pupil diameter less than 4.00mm in a dark environment
* subjects who did not cooperate well during the examination

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with simple age-related cataracts and healthy patients without systemic or eye diseases attending the Eye Optometry Hospital of Wenzhou Medical University
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional lens index | 2021.01-2021.02
  iTrace ocular aberration analyzer（itracey Technologies） to measure the preoperative DLI(Dysfunctional lens index)

SECONDARY OUTCOMES:
SS-OCT image of the lens | 2021.01-2021.02
  IOL-Master 700 biometer to measure preoperative SS-OCT image of the lens

OTHER OUTCOMES:
photos of the anterior segment | 2021.01-2021.02
  anterior segment slit lamp to take photos of the anterior segment of the subject's lens in a state of dilated pupils
self-scoring of the preoperative visual quality assessment scale | 2021.01-2021.02
  self-scoring of the preoperative Catquest-9SF visual quality assessment scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenzhou Medical University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Faria-Correia F, Ramos I, Lopes B, Monteiro T, Franqueira N, Ambrosio R Jr. Comparison of Dysfunctional Lens Index and Scheimpflug Lens Densitometry in the Evaluation of Age-Related Nuclear Cataracts. J Refract Surg. 2016 Apr;32(4):244-8. doi: 10.3928/1081597X-20160209-01. PMID 27070231
- [Background] Faria-Correia F, Ramos I, Lopes B, Monteiro T, Franqueira N, Ambrosio R Jr. Correlations of Objective Metrics for Quantifying Dysfunctional Lens Syndrome With Visual Acuity and Phacodynamics. J Refract Surg. 2017 Feb 1;33(2):79-83. doi: 10.3928/1081597X-20161206-05. PMID 28192585
- [Background] Li Z, Yu L, Chen D, Chang P, Wang D, Zhao Y, Liu S, Zhao YE. Dysfunctional Lens Index Serves as a Novel Surgery Decision-Maker for Age-Related Nuclear Cataracts. Curr Eye Res. 2019 Jul;44(7):733-738. doi: 10.1080/02713683.2019.1584676. Epub 2019 Mar 1. PMID 30822168
- See also: Dysfunctional Lens Index Serves as a Novel Surgery Decision-Maker for Age-Related Nuclear Cataracts — https://pubmed.ncbi.nlm.nih.gov/30822168/
- See also: Comparison of Dysfunctional Lens Index and Scheimpflug Lens Densitometry in the Evaluation of Age-Related Nuclear Cataracts — https://pubmed.ncbi.nlm.nih.gov/27070231/
- See also: Correlations of Objective Metrics for Quantifying Dysfunctional Lens Syndrome With Visual Acuity and Phacodynamics — https://pubmed.ncbi.nlm.nih.gov/28192585/